CLINICAL TRIAL: NCT05209867
Title: CBD-induced Biomarkers of Inflammation Reduction in People Living With HIV at the Single Cell Level
Brief Title: Single-cell CBD Biomarkers of Inflammation Reduction in People Living With HIV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Consortium for Medical Marijuana Clinical Outcomes Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB202101624 -A; OCR41346 (Other: UF OnCore)
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Results first posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Chronic Inflammation
MeSH Terms: interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- CBD Intervention (Experimental): Participants will self-administer CBD daily for 2 months.
  Interventions: Drug: CBD oil

INTERVENTIONS:
Drug: CBD oil — * Each participant will be provided two 30mL(Milliliters) bottles (2000mg CBD per bottle) with a syringe dropper during their initial (baseline) visit with instructions to administer the solution under the tongue (0.5 cc ~1/2 dropper) twice per day (BID) 8-12 hours apart (morning and evening) at the prescribed daily dosage (63mg/day).
  * The investigators plan to collect samples from five patients over three time points: baseline (no CBD), and after one and two months of CBD-administration
  Other Names: Cannabidiol

SUMMARY:
People living with HIV (PLWH) are affected by comorbidities appearing to be strongly related to chronic inflammation, a condition characterizing PLWH.

The investigators propose to study the effects of CBD on inflammation in PLWH, and establish the molecular role of different immune cells in this process. The investigators plan to use single cell RNA-sequencing (scRNAseq) to isolate CBD-specific cellular phenotypes from five persons with HIV who will provide blood samples before and after taking CBD.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to take CBD and to participate in follow up for two months
* Older than 21 and younger than 60
* Under antiretroviral therapy for 5+ years and suppressed viral load (CD4 count <350cells/ml)

Exclusion Criteria:

* Conditions/medications that may impair the immune response, e.g., rheumatoid arthritis, cancer, diabetes, chronic infections, CAD (Cold agglutinin disease), cellulitis, autoimmune diseases such as lupus, sarcoidosis
* All medications that may affect inflammation such as aspirin, steroids, statins; CD4 count <350cells/ml), pregnancy, and current marijuana or CBD use (urine drug screen)
* UF(University of Florida)/Shands staff and students will not be considered for enrollment

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simone Marini, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] Marini S, Huber A, Cash MN, Salemi M, Cook RL, Borsa P, Mavian CN. Oral Cannabidiol Treatment Is Associated with an Anti-Inflammatory Gene Expression Signature in Myeloid Cells of People Living with HIV. Cannabis Cannabinoid Res. 2024 Aug;9(4):1028-1037. doi: 10.1089/can.2023.0139. Epub 2024 Jan 22. PMID 38252549
- See also: Preprint of the study on medRxiv — https://www.medrxiv.org/content/10.1101/2023.02.24.23285761v2

RESULTS

PARTICIPANT FLOW:
Groups:
- CBD Intervention: Participants will self-administer CBD daily for 2 months.
  CBD oil: -Each participant will be provided two 30mL(Milliliters) bottles (2000mg CBD per bottle) with a syringe dropper during their initial (baseline) visit with instructions to administer the solution under the tongue (0.5 cc ~1/2 dropper) twice per day (BID) 8-12 hours apart (morning and evening) at the prescribed daily dosage (63mg/day).
  -The investigators plan to collect samples from five patients over three time points: baseline (no CBD), and after one and two months of CBD-administration
Period: Overall Study
Arm/Group | CBD Intervention
Started | 4
Completed 1 Month of Intervention (The individual completed one month of intervention and attended the second visit) | 4
Completed 2 Months of Intervention (The individual completed two months of intervention and attended the third visit) | 3
Completed | 4 (Four individuals completed the assigned intervention. One individual completed one month only. Two individuals completed two months. A fourth individual completed two months but, after protocol and data review, the quality of the provided data was deemed not sufficient (single-cell RNA was not sequenced, gene expression not measured for that individual).)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Two individuals completed the assigned intervention. A third individual completed the first month of the assigned intervention. A fourth individual completed the assigned intervention but, after review, the quality of the provided data was deemed not sufficient (single-cell RNA was not sequenced, gene expression not measured).
Arm/Group | CBD Intervention
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 2
10x single-cell gene expression [Mean (Standard Deviation); unit: Number of cells per patient] | 6553 (2111.5)
Procalcitonin [Mean (Standard Deviation); unit: NG/ML] | 0.013 (0.006)
Sedimentation Rate [Mean (Standard Deviation); unit: MM/HR] | 19 (11.3)
High-sensitivity CRP [Mean (Standard Deviation); unit: MG/L] | 4.7 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Differentially Expressed Genes
Description: Number of genes with a significant fold change before/after CBD in PBMCs (Peripheral Blood Mononuclear Cells) related to inflammation genes, calculated before and after CBD treatment (baseline and 1 month for 1 participant, 2 months for 2 participants).
Time Frame: Two time points considered: baseline, and after 1 month (1 individual) or 2 months (2 individuals)
Population: Four individuals completed the assigned intervention. One individual completed one month only. Two individuals completed two months. A fourth individual completed two months but, after protocol and data review, the quality of the provided data was deemed not sufficient (single-cell RNA was not sequenced, gene expression not measured for that individual).
Measure: Mean (Standard Deviation); unit: Differentially expressed genes
Arm/Group | CBD Intervention
Number analyzed (Participants) | 3
Differentially expressed genes | 8.3 (7)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the administration period (2 months)
Arm/Group | CBD Intervention
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBD Intervention (N=4)
Neck pain (General disorders) | 1 (1) — After the first administration of the CBD, one individual reported pain in the right side of their neck (lymph node area). Our study physician considered the neck pain likely unrelated to CBD, and safe to continue the study.

LIMITATIONS AND CAVEATS:
We processed data for individuals with different lengths of CBD exposure (2 months for two individuals; 1 month for one individual). The outcome is calculated at the single-cell level (i.e., the gene expression of each cell, from each sample, is measured), and not at the patient level. The low number of recruited patients makes impossible to draw conclusions at the patient level.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/67/NCT05209867/Prot_SAP_001.pdf